CLINICAL TRIAL: NCT05779033
Title: Ultrasound Versus Kinesiotaping in Relation to Scapular Stabilization Exercises in Shoulder Impingement Syndrome
Brief Title: Ultrasound Versus Kinesiotaping in Shoulder Impingement Syndrome
Acronym: US-SIS-KT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Heliopolis University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mohamed Kashef, B.SC physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/004362
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Impingement Syndrome
Keywords: ultrasound; kinesiotaping; Shoulder Impingement Syndrome; shoulder pain; shoulder range of motion
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Ultrasonography; Athletic Tape

STUDY DESIGN:
Intervention Model Description: Patients with shoulder impingement syndrome from both genders will participate in this study after approval of ethical committee of the faculty of physical therapy, Cairo University, and all participants provided written informed consent.
  Sample size: estimate 45 patients until we measure power analysis
  The subjects will be arranged into three groups:
  * Group I (control group) will receive scapular stabilization exercises 3 times per week for 4 weeks.
  * Group II will receive scapular stabilization exercises and Kinesiotape 3 times per week for 4 weeks.
  * Group III will receive scapular stabilization exercises and Ultrasound 3 times per week for 4 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Placebo Comparator): will receive scapular stabilization exercises 3 times per week for 4 weeks.
  Interventions: Behavioral: scapular stabilization exercises
- study group (A) (Active Comparator): will receive scapular stabilization exercises and Kinesiotape 3 times per week for 4 weeks
  Interventions: Behavioral: scapular stabilization exercises; Other: Kinesio Tape
- study group (B) (Active Comparator): will receive scapular stabilization exercises and Ultrasound 3 times per week for 4 weeks.
  Interventions: Behavioral: scapular stabilization exercises; Device: ultrasound

INTERVENTIONS:
Behavioral: scapular stabilization exercises — scapular stabilization exercises 3 times per week for 4 weeks.
Device: ultrasound — Ultrasound 3 times per week for 4 weeks.continuous US operated at a frequency of 1 MHz and at an intensity of 1.5 W/cm2 for 5 minutes
  Other Names: US
  Arms: study group (B)
Other: Kinesio Tape — Kinesiotape 3 times per week for 4 weeks. We will apply taping to two muscles (deltoideus and supraspinatus). A "Y' tape was placed over the deltoid muscle using the muscle stimulation (KT strip arms were located by stretching slightly by 15%-25%) and mechanical correction techniques (KT strip arms were located with maximal stretching). Another "Y" tape was placed over the supraspinatus muscle using the muscle inhibition technique (the starting point of the tape was attached to the sub acromial-greater tubercle with submaximal (75%) stretching and without stretching on strip arms).
  Other Names: KT
  Arms: study group (A)

SUMMARY:
studying the effect of ultrasound and kinesiotaping in shoulder impingement syndrome in reliefing pain and increase range of motion in subjects with shoulder impingement syndrome .

DETAILED DESCRIPTION:
Shoulder pain is a common presenting complaint from patients of all ages in daily clinical practice, affecting approximately one-third of individuals during their lifetime. Such pain may lead to the impairment of shoulder joint function and to severe reduction in quality of life. Shoulder impingement syndrome.

Ultrasound (US) is a physical therapy agent that is frequently used as an adjunctive treatment for shoulder pain. US has thermal and biophysical ffects which provide analgesia increases nutrition and increases blood circulation.

Kinesio taping method (KT), has been widely used also for many musculoskeletal diseases including shoulder problems. Most of taping methods are aimed to provide a mechanical stimulus for proprioception or to decrease pain by lifting skin and subcutaneous tissues.

* To investigate the effect of adding ultrasound versus Kinesiotaping to exercise program on pain intensity.
* To investigate the effect of adding ultrasound versus Kinesiotaping to exercise program on shoulder ROM.
* To investigate the effect of adding ultrasound versus Kinesiotaping to exercise program on shoulder function.
* To investigate the effect of adding ultrasound versus Kinesiotaping to exercise program on hand strength.

ELIGIBILITY:
Inclusion criteria:

1. Patients with shoulder impingement syndrome from both genders their age will be ranged and divided into three groups from 20-50 years.
2. History of shoulder pain for one month.
3. Positive Neer's impingement test and Hawkin's kiennedy test.
4. Provocation of pain above 60 degrees of flexion and abduction.

Exclusion criteria:

1. History of Shoulder girdle fracture, dislocation and surgery
2. Diagnosed with frozen shoulder or rotator cuff tear
3. History of cervicobrachial pain
4. Any neuromuscular pain in upper limb and use of corticosteroids or pain subsiding medication

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-04-09 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-08 (Actual)

PRIMARY OUTCOMES:
severity of pain | 4 weeks
  Assessed By visual analogue scale (VAS) , The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best).
Range Of Motion | 4 weeks
  assessed By Digital Goniometer
Function | 4 weeks
  assessed by disability of arm and hand quick questionnaire (quick DASH).
Hand strength | 4 weeks
  assessed by hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan hu ahmed, professor, Study Director — Cairo University
Locations (1):
- Mahmoud Ahmed Kashef, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
(age-severity of pain-range of motion function level of shoulder joint)'s of patients will be shared
Supporting Information: ICF
Time Frame: 4 weeks
Access Criteria: paper concent

REFERENCES:
- [Result] Letafatkar A, Rabiei P, Kazempour S, Alaei-Parapari S. Comparing the effects of no intervention with therapeutic exercise, and exercise with additional Kinesio tape in patients with shoulder impingement syndrome. A three-arm randomized controlled trial. Clin Rehabil. 2021 Apr;35(4):558-567. doi: 10.1177/0269215520971764. Epub 2020 Nov 6. PMID 33155484
- [Result] Gunay Ucurum S, Kaya DO, Kayali Y, Askin A, Tekindal MA. Comparison of different electrotherapy methods and exercise therapy in shoulder impingement syndrome: A prospective randomized controlled trial. Acta Orthop Traumatol Turc. 2018 Jul;52(4):249-255. doi: 10.1016/j.aott.2018.03.005. Epub 2018 Apr 25. PMID 29703659
- See also: Comparison of different electrotherapy methods and exercise therapy in shoulder impingement syndrome: A prospective randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/29703659/
- See also: Comparing the effects of no intervention with therapeutic exercise, and exercise with additional Kinesio tape in patients with shoulder impingement syndrome. A three-arm randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/33155484/